CLINICAL TRIAL: NCT06078605
Title: Efficacy of Nicotinamide on Retinal Ganglion Cell Functions in Glaucoma Patients : Clinical Trial, Cross-over Design, Double-blind, Placebo-control, Randomized, Single-center Study
Brief Title: Efficacy of Nicotinamide on Retinal Ganglion Cell Functions in Glaucoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHA University (Other)
Collaborators: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NRG1
Record Dates: First submitted 2023-02-13; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Glaucoma
Keywords: Nicotinamide; inner retinal function; retinal ganglion cell functions; Glaucoma; Vitamin B3; NAM; NRG1
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide(Mitovita) (Experimental): Group2 Baseline-6week: (Mitovita: 1.0 g/day, QD) 6-12week: (Mitovita: 2.0 g/day, BID) Crossover 12-18week: (Placebo: 1.0 g/day, QD) 18-24week: (Placebo: 2.0 g/day, BID)
  Interventions: Other: Nicotinamide(Mitovita)
- Placebo (Placebo Comparator): Group1 Baseline-6week: (Placebo: 1.0 g/day, QD) 6-12week: (Placebo: 2.0 g/day, BID) Crossover 12-18week: (Mitovita: 1.0 g/day, QD) 18-24week: (Mitovita: 2.0 g/day, BID)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Nicotinamide(Mitovita) — Nicotinamide(VitaminB3)
  Arms: Nicotinamide(Mitovita)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Efficacy of Nicotinamide on Retinal Ganglion Cell Functions in Glaucoma Patients : Clinical Trial, Cross-over Design, Double-blind, Placebo-control, Randomized, Single-center Study

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

1. Adult(Male or Female) over 19 years who were diagnosed with glaucoma.
2. In the case of participants receiving glaucoma treatment drugs, the investigator judges that the intraocular pressure remains constant for at least 1 year.
3. Intraocular pressure (IOP) >/= 8mmHg and < 18mmHg in each eye using Goldmann applanation tonometry prior to the screening visit
4. Adult participants diagnosed and treated for early-moderate glaucoma (VF mean deviation(MD) ≥-12 dB)
5. Have performed a reliable visual field in the last year, with <33% fixation losses, false positives and false negatives.
6. Written consent voluntarily to participate in this clinical trial.

Exclusion Criteria:

1. Patients with congenital glaucoma and secondary glaucoma caused by steroid drugs, etc.
2. BCVA (best-corrected visual acuity) Snellen equivalent of Snellen 20/80(logMar 0.25) or less.
3. Patients who have medical history of ocular inflammation
4. Patients with any ocular/systemic conditions that may affect electroretinogram parameter, or with visual field defects(Ischemic optic neuropathy, Proliferative diabetic retinopathy, Macular degeneration etc.)
5. Patients who have plans to intraocular surgery within the clinical trial period.
6. Patients with a history of significant ocular trauma within 6 months prior to the screening visit
7. Pregnant or lactating women.
8. A person who disagrees to contraception during a clinical trial period.
9. Patients with a history of malignancy within 5 years prior to the screening visit.
10. Patients that other researchers are determined inadequately.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of PhNR_min(photopic negative response) as measured by Electroretinogram (intra-group) | Baseline,12weeks
  Change of PhNR_min(photopic negative response) as measured by Electroretinogram after 12 weeks

SECONDARY OUTCOMES:
Change of PhNR_min(photopic negative response) as measured by Electroretinogram (intra-group) | Baseline, 6, 12, 18, 24weeks
  Change of PhNR_min(photopic negative response) as measured by Electroretinogram after 6, 12, 18 and 24 weeks
Change of PhNR_min(photopic negative response) as measured by Electroretinogram (Group1 VS Group2) | Baseline, 6, 12, 18, 24weeks
  Change of PhNR_min(photopic negative response) as measured by Electroretinogram after 6, 12, 18 and 24 weeks
Change of mean deviation as measured by Visual Fields (intra-group) | Baseline, 12weeks, 24weeks
  Change of mean deviation as measured by Visual Fields after 12 weeks and 24 weeks
Change of mean deviation as measured by Visual Fields (Group1 VS Group2) | Baseline, 12weeks, 24weeks
  Change of mean deviation as measured by Visual Fields after 12 weeks and 24 weeks
Change of Pointwise sensitivity as measured by Visual Fields (Group1 VS Group2) | Baseline, 12weeks, 24weeks
  Change of Pointwise sensitivity in glaucomatous eyes as measured by Visual Fields after 12 and 24 weeks: total/pattern deviation
Change of visual field sensitivity number of locations | Baseline, 12weeks, 24weeks
  Change of visual field sensitivity number of locations in glaucomatous eyes as measured by Visual Fields after 12 and 24 weeks: total, pattern deviation

CONTACTS AND LOCATIONS:
Overall Officials: Seungsoo Rho, MD, PhD, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- CHA University Bundang Medical Center, Seongnam, Bundang-gu, South Korea

REFERENCES:
- [Derived] Ha A, Kim YK, Lee CK, Williams PA, Morgan JE, Shin YI, Kim E, Kim M, Rho S. Effects of nicotinamide supplementation in normal-tension glaucoma: a crossover placebo-controlled randomised clinical trial. Br J Ophthalmol. 2025 Oct 30:bjo-2025-328096. doi: 10.1136/bjo-2025-328096. Online ahead of print. PMID 41167798